CLINICAL TRIAL: NCT06728436
Title: Testing the Effects of a Text Message Caregiver Support Intervention for Latinos
Acronym: CuidaTEXT R01
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH); University of Puerto Rico (Other); Icahn School of Medicine at Mount Sinai (Other); University of Miami (Other)
Responsible Party: Principal Investigator, Jaime Perales Puchalt, PhD, MPH, Assistant Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 150585; 1R01AG082306 (NIH)
Record Dates: First submitted 2024-12-06; First posted 2024-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CuidaTEXT (Experimental): 6 months of CuidaTEXT intervention + 1-month post-treatment
  Interventions: Behavioral: CuidaTEXT
- 7-Month Waitlist Control (No Intervention): Participants allocated to this arm will be offered the opportunity to start CuidaTEXT immediately after their 7 Month follow-up assessment

INTERVENTIONS:
Behavioral: CuidaTEXT — CuidaTEXT is a multidomain, bilingual 6-month text message intervention that includes delivery and content features tailored to Latino caregivers. All caregivers receive one core daily automatic message on five domains: ADRD education, social support, self-care, ADRD care management, and behavioral symptoms. Caregivers can access on-demand automatic messages to expand on the five domains via sending keywords and interact with a coach via a live chat for more personalized help.
  Arms: CuidaTEXT

SUMMARY:
The goal of this randomized clinical trial it to test the efficacy of CuidaTEXT, the first Alzheimer's disease and Related Dementias (ADRD) caregiver support intervention to capitalize on text messaging, among Latinos.

Researchers will compare those who receive the CuidaTEXT intervention to those who do not receive the intervention to see if CuidaTEXT effects Latino caregiver stressors and their negative consequences .

Participants will receive a variety of text messages, from automatic to keyword-drive, regarding ADRD education, social support, self-care, ADRD care management, and behavioral symptoms. Participants will also complete measures regarding depressive symptoms, coping, behavioral symptoms, and preparedness for caregiving.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* Spanish and English-speaking people who identify as Latino
* Reports providing hands-on care for a relative who has been given a clinical or research ADRD diagnosis and has an Eight-item Informant Interview to Differentiate Aging and Dementia (AD-8) screening score ≥2, indicating cognitive impairment
* Has a score of 7 or higher on the 10-item Center for Epidemiologic Studies Depression Scale (CESD-10)
* Self-reports being able to read and write
* Owns a cell phone with a flat fee, and uses it at least weekly for texting.

Exclusion Criteria:

* Participation in another wellbeing-related clinical trial
* Cohabitation with another participant in the CuidaTEXT R01 Study
* Participants who provide care for a person with ADRD already cared for by another participant in the CuidaTEXT R01 study
* Participant plans to move to another country within seven months

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Change in caregiver depressive symptoms | Baseline and 6 months
  Change in caregiver depressive symptoms from baseline to 6 months as measured by the 10-item Center for Epidemiologic Studies Depression Scale (CESD-10). The CES-D-10 is a self-report rating scale that measures characteristic symptoms of depression in the past week (e.g. depression, loneliness). Each item is rated on a 4-point scale (Rarely or None of the Time-Most or All of the Time). The summary score ranges from 0 to 30 with higher scores indicating higher severity.

SECONDARY OUTCOMES:
Change in caregiver behavioral distress symptoms | Baseline and 6 months
  Change in caregiver behavioral distress symptoms from baseline to 6 months as measured by the Neuropsychiatric Inventory-Questionnaire (NPI-Q).If any of 12 care recipient behavioral symptoms is present in the last month (e.g., repeating, delusions), caregivers rate their own distress on a 6-point scale (Not at All-Extreme). A distress summary score is calculated by adding the scores of all items, with scores ranging from 0 to 60. Higher scores indicate higher distress.

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Perales Puchalt, PhD, MPH, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Fairway, Kansas, United States

REFERENCES:
- [Derived] Perales-Puchalt J, Ramirez-Mantilla M, Moore HP, Velez-Uribe I, Sepulveda-Rivera V, Ruiz R, Fracachan-Cabrera M, Herrera Y, Baker C, Miras-Neira A, Bothwell B, Anderson H, Lewandowski T, Diaz FJ, Greiner KA, Williams K, Vidoni ED, Ellerbeck E, Burns JM. Testing the effects of a text message intervention on depression and distress among Latino dementia caregivers: a randomized controlled trial protocol. medRxiv [Preprint]. 2025 Sep 18:2025.09.16.25335909. doi: 10.1101/2025.09.16.25335909. PMID 41001476